CLINICAL TRIAL: NCT03083795
Title: Evaluating the Effectiveness of Social Relationships on Psychological Distress and Disease Progression in Patients With Diabetes: A Randomized Controlled Trial
Brief Title: The Effect of Social Relationships on Psychological Distress and Disease Progression in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BCDiabetes.Ca (Network)
Responsible Party: Principal Investigator, Tom Elliott, Medical Director at BC Diabetes, BCDiabetes.Ca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Love&Support
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2; Psychological Distress
Keywords: Social relationships; Vulnerable connections; Diabetes Distress; Support group
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants randomized to the social interaction cohort will meet on a monthly basis for a two hour group session designed to build social connections. In addition, participants will be paired with another study participant in this group, and will be asked to meet on a monthly basis for a minimum of 45 minutes. All participants in the social support cohort will continue to receive best standard diabetes management.
  Participants in the control group will be treated with standard diabetes care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social relationships intervention (Experimental): Participants randomized to the social interaction cohort will be split into two groups of 12. Each group of 12 will meet together once a month for a two-hour support group. Each participant will be allowed five minutes to "check-in" with the support group. During the 5 minute period the participant is encouraged to share their innermost thoughts and feelings in the knowledge that this information will not be shared outside the group.
  Participants will additionally be paired with another study participant in the same cohort and will be asked to meet outside group sessions once a week for a minimum of 45 minutes. The pairing process will take place by study investigators and will be sensitive to gender, age, and neighbourhood of residence. Participants who find that their paired partner is not suitable may ask the facilitators to help find a more suitable match.
  These participants will continue to receive BC Diabetes standard care.
  Interventions: Behavioral: Social relationships intervention
- Control cohort (No Intervention): Patients in the control group will receive BC Diabetes standard care.

INTERVENTIONS:
Behavioral: Social relationships intervention — Participants randomized to the social interaction cohort will meet on a monthly basis for a two hour group session designed to build social connections. In addition, participants will be paired with another study participant in this group, and will be asked to meet on a monthly basis for a minimum of 45 minutes. All participants in the social support cohort will continue to receive best standard diabetes management.
  Arms: Social relationships intervention

SUMMARY:
This study will determine the feasibility and effectiveness of a monthly social support group along with a weekly peer-to-peer meeting in improving perceived level of social support, diabetes distress, and A1c profiles in patients with Type II diabetes mellitus, compared with standard care offered at British Columbia Diabetes (BC Diabetes).

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded comparative group clinical trial of 48 participants receiving social interaction in addition to standard diabetes care or standard diabetes care alone. All participants will have a baseline and 6 month follow-up visit where assessment of their A1C, diabetes distress, and social support will be performed.

Participants randomized to the social interaction cohort will meet on a monthly basis for a two hour group session designed to build social connections. In addition, participants will be paired with another study participant in this group, and will be asked to meet on a monthly basis for a minimum of 45 minutes. All participants in the social support cohort will continue to receive best standard diabetes management.

Participants in the control group will be treated with standard diabetes care. At the end of the 6-month study, they will have the opportunity to engage in the same social interventions offered to the social interaction group.

ELIGIBILITY:
Inclusion Criteria:

* Willingly provide your full informed consent to participate;
* Are at least 19 years of age;
* Have an established diagnosis of Type 2 diabetes mellitus;
* Have a Diabetes Distress Screening Scale (a score of 2-3 is considered moderate distress, 3-4 is considered high)
* Have a Social Provisions Scale score less than 60 (a score of 80-90 is considered high, 60-80 moderate and less than 60 sub-optimal)
* Have an A1c greater than 8.5% in the last 2 months (a score of 6-7 is considered optimal, 7-8 sub-optimal and >8.0 inadequate)

Exclusion Criteria:

* Are unable to easily communicate in oral and written English.
* Have a physical disability or psychiatric diagnosis which would limit the ability to participate in the study;
* Are a prisoner, or in pre-trial;
* Do not have a fixed address;

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
A1C | 6 months post randomization
  Hemoglobin A1C blood test
Diabetes distress | 6 months post randomization
  Score on Diabetes Distress Screening Scale
Self-reported social support | 6 months post randomization
  Score on Social Provisions Scale

SECONDARY OUTCOMES:
Blood pressure | 6 months post randomization
  Blood pressure
Medical adherence | 6 months post randomization
  Participants will indicate their level of medication adherence on a scale of 1-5. To do this, they will respond to the question "To what extent do you agree with the following statement: I reliably take my diabetes-related medication", where the possible responses are: strongly disagree, disagree, neutral, agree, strongly agree. These responses will be converted into a 5-point scale where strongly disagree = 1 and strongly agree = 5
Statin refusal | 6 months post randomization
  Participants will score yes (if they refuse statin treatment) or no (if they do not refuse statin treatment)
Diet | 6 months post randomization
  Participants will score their diet on a scale of 1-5. To do this, they will respond to the question " I currently have a good diet", where the possible responses are: strongly disagree, disagree, neutral, agree, strongly agree. These responses will be converted into a 5-point scale where strongly disagree = 1 and strongly agree = 5
Exercise | 6 months post randomization
  Participants will score their exercise on a scale of 1-5. To do this, they will respond to the question "I currently get enough exercise", where the possible responses are: strongly disagree, disagree, neutral, agree, strongly agree. These responses will be converted into a 5-point scale where strongly disagree = 1 and strongly agree = 5
Weight | 6 months post randomization
  Weight will be recorded in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elliott, MBBS, Principal Investigator — BC Diabetes, The University of British Columbia

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the study, anonymized participant data may be shared with other researchers wishing to undergo similar studies to assist with study design and implementation.

REFERENCES:
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Byrne D, Alvaregna M editors. Handbook of Psychocardiology. 1st ed. New York: Springer; 2016.
- [Background] Ducat L, Philipson LH, Anderson BJ. The mental health comorbidities of diabetes. JAMA. 2014 Aug 20;312(7):691-2. doi: 10.1001/jama.2014.8040. No abstract available. PMID 25010529
- [Background] Feng X, Astell-Burt T. What types of social interactions reduce the risk of psychological distress? Fixed effects longitudinal analysis of a cohort of 30,271 middle-to-older aged Australians. J Affect Disord. 2016 Nov 1;204:99-102. doi: 10.1016/j.jad.2016.06.041. Epub 2016 Jun 14. PMID 27344617
- [Background] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Background] Hackett RA, Steptoe A. Psychosocial Factors in Diabetes and Cardiovascular Risk. Curr Cardiol Rep. 2016 Oct;18(10):95. doi: 10.1007/s11886-016-0771-4. PMID 27566328
- [Background] Ismail K, Winkley K, Rabe-Hesketh S. Systematic review and meta-analysis of randomised controlled trials of psychological interventions to improve glycaemic control in patients with type 2 diabetes. Lancet. 2004 May 15;363(9421):1589-97. doi: 10.1016/S0140-6736(04)16202-8. PMID 15145632
- [Background] Rabi DM, Edwards AL, Southern DA, Svenson LW, Sargious PM, Norton P, Larsen ET, Ghali WA. Association of socio-economic status with diabetes prevalence and utilization of diabetes care services. BMC Health Serv Res. 2006 Oct 3;6:124. doi: 10.1186/1472-6963-6-124. PMID 17018153
- [Background] O'Kane C, O'Kane D. Real: The Power of Authentic Connection. 1st ed. Clearmind publishing; 2016.
- [Background] Rossi MC, Lucisano G, Funnell M, Pintaudi B, Bulotta A, Gentile S, Scardapane M, Skovlund SE, Vespasiani G, Nicolucci A; BENCH-D Study Group. Interplay among patient empowerment and clinical and person-centered outcomes in type 2 diabetes. The BENCH-D study. Patient Educ Couns. 2015 Sep;98(9):1142-9. doi: 10.1016/j.pec.2015.05.012. Epub 2015 May 21. PMID 26049679
- [Background] Siousioura D. Review of therapeutic groups for type 1 diabetes mellitus patients. J Endocrinol Diabetes 2012;3(2):11-21.
- [Background] Young-Hyman D, de Groot M, Hill-Briggs F, Gonzalez JS, Hood K, Peyrot M. Erratum. Psychosocial Care for People With Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care 2016;39:2126-2140. Diabetes Care. 2017 Feb;40(2):287. doi: 10.2337/dc17-er02. Epub 2016 Dec 7. No abstract available. PMID 27927693